CLINICAL TRIAL: NCT02656069
Title: G-Pen (Glucagon Injection) Compared to Lilly Glucagon (Glucagon for Injection [RDNA Origin]) for Induced Hypoglycemia Rescue in Adult Patients With T1DM: A Phase 3, Multi-center, Randomized, Blinded, 2-Way Crossover Study to Evaluate Efficacy and Safety
Brief Title: Safety and Efficacy of G-Pen Compared to Lilly Glucagon for Hypoglycemia Rescue in Adult Type 1 Diabetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xeris Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: XSGP-301
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Results first posted 2018-09-28 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-09

CONDITIONS: Hypoglycemia; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1 | interventions — Glucagon

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- G-Pen first, then Lilly Glucagon (Other): A single 1 mg subcutaneous (SC) injection of G-Pen (glucagon injection) with a 7-28 day wash-out, followed by a single 1 mg SC injection of Lilly Glucagon (glucagon injection [rDNA origin])
  Interventions: Drug: G-Pen (glucagon injection); Drug: Lilly Glucagon (glucagon injection [rDNA origin])
- Lilly Glucagon first, then G-Pen (Other): A single 1 mg SC injection of Lilly Glucagon (glucagon injection [rDNA origin]) with a 7-28 day wash-out, followed by a single 1 mg SC injection of G-Pen (glucagon injection)
  Interventions: Drug: G-Pen (glucagon injection); Drug: Lilly Glucagon (glucagon injection [rDNA origin])

INTERVENTIONS:
Drug: G-Pen (glucagon injection) — 1 mg of pre-mixed liquid Xeris glucagon delivered via auto-injector
  Other Names: glucagon
Drug: Lilly Glucagon (glucagon injection [rDNA origin]) — 1 mg of Lilly glucagon reconstituted from lyophilized powder
  Other Names: glucagon

SUMMARY:
This is a blinded, randomized crossover study to compare the safety and efficacy of G-Pen (glucagon injection) to Lilly Glucagon (glucagon for injection [rDNA origin]) for hypoglycemia rescue of adult patients with type 1 diabetes.

DETAILED DESCRIPTION:
This is a blinded, randomized, Phase 3 comparative efficacy and safety study in adults with type 1 diabetes. Patients will complete screening procedures up to 60 days before randomization to determine eligibility before enrollment to the treatment phase.

The procedure for evaluating the efficacy of the G-Pen (glucagon injection) consists of inducing hypoglycemia by intravenous administration of regular insulin diluted in normal saline. Each participant will undergo two episodes of insulin-induced hypoglycemia, and in random order will receive 1 mg G-Pen (glucagon injection) during one episode and 1 mg Lilly Glucagon during the other episode. There will be wash out period of 7-28 days between treatment visits.

Blood glucose levels will be monitored post-dosing, with a return of plasma glucose to a concentration > 70 mg/dL within 30 minutes signifying successful hypoglycemia rescue. As a confirmation of efficacy, subjects will complete a questionnaire concerning changes in symptoms of hypoglycemia following treatment with glucagon.

Subjects will return for a follow-up safety visit 3-14 days following administration of the final dose of glucagon.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 1 diabetes mellitus for at least 24 months
* usage of daily insulin treatment
* random serum C-peptide concentration < 0.5 ng/mL

Exclusion Criteria:

* pregnant or nursing
* HbA1c >9.0%
* renal insufficiency
* hepatic synthetic insufficiency
* aspartate or alanine aminotransferase > 3 times the upper limit of normal
* hematocrit less than or equal to 30%
* use of > 2.0 U/kg total insulin dose per day
* inadequate bilateral venous access in both arms
* congestive heart failure, New York Heart Association class II, III or IV
* active malignancy within 5 years, except basal cell or squamous cell skin cancers
* history of breast cancer or malignant melanoma
* major surgical operation within 30 days
* current seizure disorder.
* current bleeding disorder, treatment with warfarin, or platelet count below 50,000
* history of pheochromocytoma or disorder with increased risk of pheochromocytoma
* history of insulinoma
* history of glycogen storage disease.
* positive for HIV, hepatitis C virus or active hepatitis B virus infection
* whole blood donation of 1 pint (500 mL) within 8 weeks
* active substance or alcohol abuse
* administration of glucagon within 28 days
* participation in other studies involving an investigational drug or device within 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-09-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - ProSciento, Inc., Chula Vista, California
  - AMCR Institute, Escondido, California
  - Diablo Clinical Research, Walnut Creek, California
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Rainier Research, Renton, Washington
- LMC Diabetes & Endocrinology, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christiansen MP, Cummins M, Prestrelski S, Close NC, Nguyen A, Junaidi K. Comparison of a ready-to-use liquid glucagon injection administered by autoinjector to glucagon emergency kit for the symptomatic relief of severe hypoglycemia: two randomized crossover non-inferiority studies. BMJ Open Diabetes Res Care. 2021 Oct;9(1):e002137. doi: 10.1136/bmjdrc-2021-002137. PMID 34620618

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period began 15 March 2017 and ran through 30 June 2017. Subjects were screened for study eligibility at one of the 7 clinical sites up to 60 days prior to randomization.
Pre-assignment Details: A total of 6 screened and eligible subjects were not randomized to one of the treatment sequences due to closing of the enrollment period.
Groups:
- G-Pen First, Then Lilly Glucagon: A single 1 mg subcutaneous (SC) injection of G-Pen™ (glucagon injection) with a 7-28 day wash-out, followed by a single 1 mg SC injection of Lilly Glucagon (glucagon injection [rDNA origin])
  G-Pen™ (glucagon injection): 1 mg of pre-mixed liquid Xeris glucagon delivered via auto-injector
  Lilly Glucagon (glucagon injection [rDNA origin]): 1 mg of Lilly glucagon reconstituted from lyophilized powder
- Lilly Glucagon First, Then G-Pen: A single 1 mg SC injection of Lilly Glucagon (glucagon injection [rDNA origin]) with a 7-28 day wash-out, followed by a single 1 mg SC injection of G-Pen™ (glucagon injection)
  Lilly Glucagon (glucagon injection [rDNA origin]): 1 mg of Lilly glucagon reconstituted from lyophilized powder
  G-Pen™ (glucagon injection): 1 mg of pre-mixed liquid Xeris glucagon delivered via auto-injector
Period: First Intervention
Arm/Group | G-Pen First, Then Lilly Glucagon | Lilly Glucagon First, Then G-Pen
Started | 44 | 36
Completed | 44 | 36
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | G-Pen First, Then Lilly Glucagon | Lilly Glucagon First, Then G-Pen
Started | 44 | 36
Completed | 43 | 35
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: All eligible, randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | G-Pen First, Then Lilly Glucagon | Lilly Glucagon First, Then G-Pen | Total
Number analyzed (Participants) | 44 | 36 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 31 | 71
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (15.55) | 45.5 (14.87) | 43.6 (15.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 29 | 21 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic White | 38 | 29 | 67
  Race/Ethnicity: Hispanic | 2 | 4 | 6
  Race/Ethnicity: African American | 2 | 2 | 4
  Race/Ethnicity: Other | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  North America: Canada | 4 | 4 | 8
  North America: United Staates | 40 | 32 | 72

OUTCOME MEASURES:

1. Primary Outcome: Hypoglycemia Rescue: Intent-to-Treat Population
Description: Number of subjects with an increase in plasma glucose concentration from below 50 mg/dL to greater than 70 mg/dL within 30 minutes after administration of glucagon
Time Frame: At 30 minutes following administration of study drug
Population: Modified intent-to-treat population of all randomized subjects analyzed by actual treatment received
Measure: Count of Participants; unit: Participants
Groups:
- G-Pen: A single 1 mg subcutaneous (SC) injection of G-Pen™ (glucagon injection)
- Lilly Glucagon: A single 1 mg subcutaneous (SC) injection of Lilly Glucagon
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 78 | 79
Participants | 74 | 79

2. Primary Outcome: Hypoglycemia Rescue: Per Protocol Population
Description: as for outcome 1
Time Frame: At 30 minutes following administration of study drug
Population: All randomized, treated subjects without a major protocol violation
Measure: Count of Participants; unit: Participants
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 77 | 78
Participants | 74 | 78

3. Primary Outcome: Hypoglycemia Rescue: Alternate Glucose Response Definition
Description: Number of subjects with either an increase in plasma glucose concentration from below 50 mg/dL to greater than 70 mg/dL or an increase in from baseline in plasma glucose concentration of at least 20 mg/dL within 30 minutes after administration of glucagon
Time Frame: At 30 minutes following administration of study drug
Population: Modified intent-to-treat population of all randomized subjects analyzed by actual treatment received
Measure: Count of Participants; unit: Participants
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 78 | 79
Participants | 76 | 79

4. Secondary Outcome: Plasma Glucose Area Under the Curve (AUC)
Description: Pharmacodynamic endpoint of plasma glucose AUC from baseline to 90 minutes following administration of glucagon
Time Frame: At -5, 0, 10, 20, 30, 45, 60, and 90 minutes following administration of glucagon
Population: Modified intent-to-treat population of all randomized subjects analyzed by actual treatment received
Measure: Mean (Standard Deviation); unit: mg*min/dL
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 78 | 79
mg*min/dL | 11651.4 (2406.9) | 12260.4 (2134.2)

5. Secondary Outcome: Plasma Glucose Maximum Concentration (Cmax)
Description: Pharmacodynamic endpoint of plasma glucose Cmax from baseline to 4 hours following administration of glucagon
Time Frame: At -5, 0, 10, 20, 30, 45, 60, 90, 120, 180 and 240 minutes following administration of glucagon
Population: Modified intent-to-treat population of all randomized subjects analyzed by actual treatment received
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 78 | 79
mg/dL | 202.7 (41.8) | 193.5 (42.2)

6. Secondary Outcome: Plasma Glucose Time to Maximum Concentration (Tmax)
Description: Pharmacodynamic endpoint of plasma glucose Tmax from baseline to 4 hours following administration of glucagon
Time Frame: At -5, 0, 10, 20, 30, 45, 60, 90, 120, 180 and 240 minutes following administration of glucagon
Population: Modified intent-to-treat population of all randomized subjects analyzed by actual treatment received
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 78 | 79
minutes | 111.3 (33.5) | 100.4 (42.7)

7. Secondary Outcome: Plasma Glucose Time to Concentration > 70 mg/dL
Description: Pharmacodynamic endpoint of time to achieve a plasma glucose concentration > 70 mg/dL following administration of glucagon
Time Frame: At -5, 0, 10, 20, 30, 45, 60, 90, 120, 180 and 240 minutes following administration of glucagon
Population: Modified intent-to-treat population of all randomized subjects analyzed by actual treatment received
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 78 | 79
minutes | 19.9 (8.5) | 14.2 (4.3)

8. Secondary Outcome: Time to Resolution of Hypoglycemia Symptoms
Description: Time to resolution of mean autonomic, mean neuroglycopenic and mean total hypoglycemia symptom scores from baseline through 90 minutes following administration of glucagon.
Time Frame: At 0, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 65, 70, 75, 80, 85 and 90 minutes following administration of glucagon
Population: Modified intent-to-treat population of all randomized subjects analyzed by actual treatment received
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 77 | 79
minutes
  Autonomic Symptoms | 16.0 (11.5) | 14.2 (9.4)
  Neuroglycopenic Symptoms | 16.7 (10.2) | 14.3 (9.0)
  All Symptoms | 19.8 (11.7) | 17.0 (8.9)

9. Secondary Outcome: Global Assessment of Hypoglycemia
Description: Time to resolution of the overall sensation of hypoglycemia following administration of glucagon
Time Frame: as for outcome 8
Population: Modified intent-to-treat population of all randomized subjects analyzed by actual treatment received
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 76 | 79
minutes | 16.8 (10.7) | 15.7 (8.3)

10. Post Hoc Outcome: Hypoglycemia Rescue: Glucose or Symptomatic Response Definition
Description: Number of subjects with either an increase in plasma glucose concentration from below 50 mg/dL to greater than 70 mg/dL or resolution of all neuroglycopenic symptoms of hypoglycemia within 30 minutes after administration of glucagon
Time Frame: At 30 minutes following administration of study drug
Population: Modified intent-to-treat population of all randomized subjects analyzed by actual treatment received
Measure: Count of Participants; unit: Participants
Arm/Group | G-Pen | Lilly Glucagon
Number analyzed (Participants) | 78 | 79
Participants | 78 | 79

ADVERSE EVENTS:
Time Frame: For the first intervention, treatment emergent adverse events were defined as adverse events occurring at any time after receipt of the first intervention and prior to receipt of the second intervention, 7-28 days later. For the second intervention, treatment emergent adverse events were defined as adverse events occurring at any time after receipt of the second intervention and prior to completion of the follow-up evaluation visit occurring 3-14 days later.
Arm/Group | G-Pen | Lilly Glucagon
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/78 | 1/79
Other Adverse Events (participants affected / at risk) | 24/78 | 16/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-Pen (N=78) | Lilly Glucagon (N=79)
hyperinsulinemic hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1) — The evening after receiving Lilly Glucagon 1 mg, a subject had severe hypoglycemia at home requiring 3rd party assistance. An emergency medical technician administered saline. The subject recovered with no sequelae and completed the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-Pen (N=78) | Lilly Glucagon (N=79)
Nausea (Gastrointestinal disorders) | 17 (18) | 10 (10)
Vomiting (Gastrointestinal disorders) | 5 (5) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT02656069/Prot_SAP_000.pdf